CLINICAL TRIAL: NCT07012928
Title: Local Clinical and Immunological Responses in Eosinophilic Esophagitis (EoE) Patients, Role of Mucosal Barrier Function and Type II Inflammation
Acronym: SINFONIA
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof.dr. A.J. (Arjan) Bredenoord, Prof. Dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: 2024.0849; Sanofi (Other Grant/Funding Number: Sanofi Pathways in Type 2 Inflammation Global Innovation Grant)
Record Dates: First submitted 2025-05-15; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Eosinophilic Esophagitis (EoE)
Keywords: Eosinophilic Esophagitis; Dupilumab; Permeability esophagus; TEER
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and esophagus biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Dupilumab: Blood, biopsies, questionnaire
- Active EoE disease: Blood, biopsies, questionnaire
- Control: Blood, biopsies

SUMMARY:
Eosinophilic esophagitis (EoE) is an allergic inflammation of the esophagus. If not treated properly, inflammation and narrowing of the esophagus can occur. This can eventually lead to food impaction. Food allergens play an important role in the pathogenesis of EoE, as demonstrated by endoscopic and clinical resolution of EoE once the causative food is removed from the diet and exacerbation when the same food is reintroduced Similarly, amino acid-based

elemental diets are effective in both adults and children with EoE. However, the exact mechanism by which food allergens can initiate inflammation in EoE is still unknown, as there are limited data on the early local esophageal immune response after challenge with a specific food trigger. Previous research has shown that this can be treated with antacids (PPI) and corticosteroids. This reduces the permeability of the esophagus (which is increased in EoE), but not to the level of healthy individuals. Most likely this is due to a mild underlying allergic inflammation that persists under treatment with the above agents. The idea is that dupilumab inhibits this type II inflammation, which will further reduce the permeability. In addition, the effect of food allergens on esophageal biopsies from both EoE patients and healthy patients will be examined. This will then be compared to the biopsies taken after the use of dupilumab.

ELIGIBILITY:
Inclusion Criteria:

EoE patient group with dupilumab or topical budesonide Previous diagnosis of active EoE confirmed by histopathology e.g. presence of 15 or more eosinophilic granulocytes per hpf in mid or proximal esophageal biopsies Scheduled to start with dupilumab or topical budesonide as regular care 18 to 75 years of age Written informed consent must be obtained and documented

EoE patient group with active EoE Previous diagnosis of active EoE confirmed by histopathology e.g. presence of 15 or more eosinophilic granulocytes per hpf in mid or proximal esophageal biopsies Scheduled for an upper endoscopy 18 to 75 years of age Written informed consent must be obtained and documented

Non-EoE control group Scheduled for a upper endoscopy for other, non-esophageal related, symptoms 18 to 75 years of age Written informed consent must be obtained and documented

Exclusion Criteria:

EoE patient group with dupilumab, topical budesonide and with active EoE Use of oral or systemic antihistaminics, oral cromoglicates, systemic corticosteroids, leukotriene inhibitors or monoclonal antibodies, in the month preceding the study Proven gastroesophageal reflux disease or other cause for esophageal eosinophilia, History of peptic ulcer disease, History of Barrett's esophagus, History of gastro intestinal cancer or ASA class III, IV or V

Non-EoE control group Symptoms suggestive of esophageal disease or other disease that may infolve the esophagus Personal history of atopic, skin or systemic diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Most of the patients will have active EoE at the beginning, 12 will be treated with dupilumab, 20 active disease patients. There will be 12 patients without EoE
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Local clinical and immunological responses in eosinophilic esophagitis (EoE) patients, role of mucosal barrier function and type II inflammation | 26 weeks after dupilumab
  Esophagael barrier function improvement after 26 week of dupilumab treatment in EoE patients, assessed by the change in transepithelial electrical resistance (TEER).

SECONDARY OUTCOMES:
Food-induced immune responses in EoE patients after dupilumab | 26 weeks after dupilumab
  food-induced immune responses in esophageal biopsy specimens exposed to different food allergens ex vivo after dupilumab.

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Depends on the results